CLINICAL TRIAL: NCT02605512
Title: Early Detection and Prediction of Cardiotoxicity in Radiotherapy-treated Breast Cancer Patients
Brief Title: BreAst Cancer and Cardiotoxicity Induced by RAdioTherapy: the BACCARAT Study
Acronym: BACCARAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sophie JACOB (Other Government)
Collaborators: Institut de Radioprotection et de Surete Nucleaire (Other Government); Clinique Pasteur (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor-Investigator, Sophie JACOB, PhD, Institut de Radioprotection et de Surete Nucleaire
Organization: Institut de Radioprotection et de Surete Nucleaire (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRSN_2015-A00990-49
Record Dates: First submitted 2015-11-06; First posted 2015-11-16 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Cardiac Toxicity
Keywords: Radiotherapy; Echocardiography; Strain strain rate; Coronary computed tomography angiography; Segments of coronary arteries; Subclinical functional and anatomical cardiac lesions; Biomarkers; Heart dosimetry
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breast cancer patients with 3DCRT (Other): Measures of subclinical functional and anatomical cardiac lesions and circulating biomarkers 'Subclinical cardiac lesions and biomarkers'
  Interventions: Other: Subclinical cardiac lesions and biomarkers

INTERVENTIONS:
Other: Subclinical cardiac lesions and biomarkers — Functional myocardial dysfunction based on 2D-speckle tracking echocardiography, Anatomical coronary lesions based on Coronary computed tomography angiography, a panel of circulating biomarkers based on blood samples and plasma

SUMMARY:
Breast radiotherapy RT used until the 1990s was clearly responsible for increased mortality due to long term cardiac complications. Since the 2000s, improvements have appeared in dose distributions to organ at risks such as heart, but now, little is known on the risk of potential cardiac impairment in this population, in particular for chemotherapy naive patients. Based on the state that clinically detectable cardiotoxicity is generally preceded by subclinical cardiac dysfunctions, the aim of the BACCARAT study (BreAst Cancer and Cardiotoxicity induced by RAdioTherapy) is to evaluate whether adjuvant 3DCRT induces cardiac toxicity that could be detected in the first two years after treatment based on a global approach with repeated analysis of subclinical functional and anatomical cardiac lesions in myocardial and coronary levels and circulating biomarkers.

DETAILED DESCRIPTION:
BACCARAT study consists in a monocentric prospective cohort study that will finally include 120 women treated with adjuvant RT for breast cancer in the Clinique Pasteur in Toulouse, and followed for 2 years after RT.

Women aged 50 to 70 years, treated for breast cancer and for whom adjuvant 3DCRT is indicated, without chemotherapy are eligible for the study.

Baseline and follow-up include measures of functional myocardial dysfunction based on 2D-speckle tracking echocardiography, anatomical coronary lesions based on Coronary computed tomography angiography, and a wide panel of circulating biomarkers. Absorbed doses is evaluated for whole heart and for each different parts of heart, in particular coronary arteries.

Analysis on occurrence and evolutions of subclinical cardiac lesions and biomarkers will be performed and completed with dose-response relations with absorbed doses of different heart segments.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 70 years
* Women surgically treated for left or right breast cancer and for whom adjuvant treatment is radiotherapy with irradiation of the breast or chest wall irradiation and possibly ganglion chains,
* Adjuvant radiotherapy with 3DCRT performed in Clinique Pasteur Toulouse
* WHO performance status ECOG - Eastern Cooperative Oncology Group (index normally used to describe the patient's condition) = 0 or 1
* Being volunteer to participate in the study and have signed the consent form

Exclusion Criteria:

* Indication of adjuvant chemotherapy
* Clinically or radiologically detectable metastasis
* Personal history of coronary artery disease or myocardial disease
* Personal history of breast cancer or other cancer requiring radiotherapy to the thorax
* Patient with controlled infection or severe disease and / or non-hazardous to their participation in the study
* Contraindications to injection of iodinated contrast (for CCTA): pregnancy, renal failure, allergy.
* Pregnancy, lactation
* Abnormal echocardiography before radiotherapy:
* LVEF <50%
* Longitudinal strain> - 16%
* Longitudinal strain rate <1% / s
* Abnormal wall motion
* CCTA before radiotherapy showing that therapeutic management is required (coronary-artery calcium (CAC) score>600)

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with decreased myocardial function assessed by echocardiography | 2 years after 3DCRT (baseline measures performed before radiotherapy)
  Number of patients with a decrease in the mean strain or strain rate measured from the echocardiography of the order of 5% between the measurement before RT and 24 months after RT
Number of patients with increased coronary plaques assessed by CT coronary angiography | 2 years after 3DCRT (baseline measures performed before radiotherapy)
  Number of patients with an increase of the average index of coronary plaques measured from the CT coronary angiography in the order of 15% between the measurements before RT and 24 months after RT

SECONDARY OUTCOMES:
Decrease in the strain or strain rate | 6 months after 3DCRTand 2 years after 3DCRT (baseline measures performed before radiotherapy)
Modification in series of circulating biomarkers of cardiac lesions | 5 weeks after initiation of 3DCRT (corresponding to the end of 3DCRT sessions), 6 months after 3DCRTand 2 years after 3DCRT (baseline measures performed before radiotherapy)
  Classical biomarkers of cardiac injury: C-reactive protein, Troponin I, B-type natriuretic peptide (NT-Pro BNP), beta2-Microglobulin, Galectin 3 / Inflammatory cytokines: Interleukin 6, Interleukin 8, Interleukin 18, TNF-α / Endothelial activation and dysfunction: sVCAM,-1 , s-ICAM-1, E-selectin, P-selectin , vWF, PAI-1, Fibrinogen , Thrombomodulin, TGF-β1 / Microparticles: CD14, CD31, CD41, CD3, CD235a / microRNAs : miR-1, miR-133, miR-208, miR-499, miR-126, miR-130, miR-145, miR-181, miR-150, miR-155, miR-223, miR-17, miR-18, miR-22, miR-34, miR-92, miR-140, miR-182, miR-199, miR-423, miR-590
Correlation between the absorbed radiation dose by the whole heart and different structures of the heart and measurements of strain and strain rate and indices of coronary plaques | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Atul Pathak, MD PhD, Principal Investigator — Clinique Pasteur Toulouse
Locations (1):
- Clinique Pasteur, Toulouse, France

REFERENCES:
- [Derived] Honaryar MK, Locquet M, Allodji R, Jimenez G, Pinel B, Lairez O, Panh L, Camilleri J, Broggio D, Ferrieres J, De Vathaire F, Jacob S. Cancer therapy-related cardiac dysfunction after radiation therapy for breast cancer: results from the BACCARAT cohort study. Cardiooncology. 2024 Aug 26;10(1):54. doi: 10.1186/s40959-024-00255-9. PMID 39187877
- [Derived] Honaryar MK, Allodji R, Jimenez G, Lapeyre M, Panh L, Camilleri J, Broggio D, Ferrieres J, De Vathaire F, Jacob S. Early Development of Atherosclerotic Plaques in the Coronary Arteries after Radiotherapy for Breast Cancer (BACCARAT Study). J Cardiovasc Dev Dis. 2023 Jul 12;10(7):299. doi: 10.3390/jcdd10070299. PMID 37504555
- [Derived] Walker V, Lairez O, Fondard O, Jimenez G, Camilleri J, Panh L, Broggio D, Bernier MO, Laurier D, Ferrieres J, Jacob S. Myocardial deformation after radiotherapy: a layer-specific and territorial longitudinal strain analysis in a cohort of left-sided breast cancer patients (BACCARAT study). Radiat Oncol. 2020 Aug 20;15(1):201. doi: 10.1186/s13014-020-01635-y. PMID 32819449
- [Derived] Walker V, Lairez O, Fondard O, Pathak A, Pinel B, Chevelle C, Franck D, Jimenez G, Camilleri J, Panh L, Broggio D, Derreumaux S, Bernier MO, Laurier D, Ferrieres J, Jacob S. Early detection of subclinical left ventricular dysfunction after breast cancer radiation therapy using speckle-tracking echocardiography: association between cardiac exposure and longitudinal strain reduction (BACCARAT study). Radiat Oncol. 2019 Nov 14;14(1):204. doi: 10.1186/s13014-019-1408-8. PMID 31727075
- [Derived] Jacob S, Camilleri J, Derreumaux S, Walker V, Lairez O, Lapeyre M, Bruguiere E, Pathak A, Bernier MO, Laurier D, Ferrieres J, Gallocher O, Latorzeff I, Pinel B, Franck D, Chevelle C, Jimenez G, Broggio D. Is mean heart dose a relevant surrogate parameter of left ventricle and coronary arteries exposure during breast cancer radiotherapy: a dosimetric evaluation based on individually-determined radiation dose (BACCARAT study). Radiat Oncol. 2019 Feb 7;14(1):29. doi: 10.1186/s13014-019-1234-z. PMID 30732640
- [Derived] Jacob S, Pathak A, Franck D, Latorzeff I, Jimenez G, Fondard O, Lapeyre M, Colombier D, Bruguiere E, Lairez O, Fontenel B, Milliat F, Tamarat R, Broggio D, Derreumaux S, Ducassou M, Ferrieres J, Laurier D, Benderitter M, Bernier MO. Early detection and prediction of cardiotoxicity after radiation therapy for breast cancer: the BACCARAT prospective cohort study. Radiat Oncol. 2016 Apr 7;11:54. doi: 10.1186/s13014-016-0627-5. PMID 27056179